CLINICAL TRIAL: NCT06832046
Title: Evaluation of the "Intranasal Fentanyl" Protocol in Pediatric Surgical Emergencies at Strasbourg University Hospital
Acronym: TraumaDol
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9480
Record Dates: First submitted 2025-02-10; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Pain
Keywords: Pain Syndrome; Intranasal Fentanyl; pediatric; Pediatric surgical emergency
MeSH Terms: conditions — Musculoskeletal Pain; Somatoform Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency trauma departments receive thousands of patients each year whose main symptom is pain. In recent years, intranasal fentanyl (FIN) has entered the therapeutic arsenal to treat pain in the emergency department. Various studies have validated its effectiveness for musculoskeletal pain as well as its tolerance and safety of use. Since then, new protocols have been implemented including this treatment. In This study, the investigators propose to retrospectively study the quality of prescription of intranasal fentanyl in the treatment of pain in the emergency department and the quality of monitoring of this treatment in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Child < 18 years old
* Child treated in the pediatric emergency department of Strasbourg University Hospital
* Child who has benefited from intranasal fentanyl between 08/01/2022 and 09/31/2024.
* Child (and/or his/her parental authority) who has not expressed, after information, his/her (their) opposition to the reuse of his/her health data for the purposes of this research.

Exclusion Criteria:

* Refusal of the child (and/or his/her parent) to participate in the study
* Patient's medical file not incomplete
* Child not domiciled in France.

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Child < 18 years old who has benefited from intranasal fentanyl between 08/01/2022 and 09/31/2024.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
The judgment criterion is composite in order to retrospectively evaluate the relevance of the prescription, administration and monitoring of the intranasal fentanyl (FIN) protocol. | Up to 2 years
  The judgment criterion includes, 1) the prescription and 2) the administration and monitoring.
  1) Concerning the prescription:
  * Compliance with the contraindications of intranasal fentanyl (weight less than 10kg and/or age less than 1 year).
  * Compliance with the medical indication according to the protocol (pathologies and/or procedures performed and/or initial assessment of pain).
  * Compliance with the prescription terms (indication of the dead space, unit, route of administration and dose).
The judgment criterion is composite in order to retrospectively evaluate the relevance of the prescription, administration and monitoring of the intranasal fentanyl (FIN) protocol.The judgment criterion includes, | Up to 2 years
  The judgment criterion includes, 1) the prescription and 2) the administration and monitoring.
  2) Concerning the administration and monitoring:
  * Compliance with the double nursing check, product administration schedule and identification of the caregiver.
  * Nursing monitoring in accordance with the protocol, i.e. taking hemodynamic and respiratory constants (Sat02, FR, FC and TA) before taking fentanyl, at 10-15 minutes, at 30 minutes and at 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urgences Médico-Chirurgicales Pédiatriques - CHU de Strasbourg - France, Strasbourg, France